CLINICAL TRIAL: NCT01883375
Title: Dignity Talk: a Novel Palliative Care Intervention for Patients and Their Families
Brief Title: Dignity Talk: Helping Palliative Care Patients and Families Have Important Conversations
Acronym: DTalk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: H2013:024
Record Dates: First submitted 2013-02-11; First posted 2013-06-21 (Estimated); Last update posted 2017-12-14 (Actual); Status verified 2016-11

CONDITIONS: Palliative Care; Family; End of Life Care
Keywords: Palliative Care; Family; adaptation, psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dignity Talk dyad completers (Experimental): Those dyads where both patient and family member co-participant complete the protocol using the Dignity Talk Communication Topics
  Interventions: Behavioral: Dignity Talk
- Dignity Talk non-completers (Experimental): Those dyads where patient and family member co-participant either do not complete the protocol or do not use the Dignity Talk Communication Topics (November 2016 - the investigators have not as yet enrolled any participants who have not completed the study without using the Dignity Talk Topics. However some participants have withdrawn from the study without completing.
  Interventions: Behavioral: The Dignity Talk Communication Topics

INTERVENTIONS:
Behavioral: Dignity Talk — Patient and family member participants will be given the Dignity Talk framework questions and asked to use them in conversation with each other. Research nurse will return at day 4-6 to confirm both participants have covered all items they wish to discuss. 4-6 months after the death of patient, family members will be contacted in order to collect data pertaining to their bereavement experiences and distress. Will also be asked to complete evaluative feedback on Dignity Talk.
  Arms: Dignity Talk dyad completers
Behavioral: The Dignity Talk Communication Topics — There have not been any non-completers - this arm not being used currently
  Arms: Dignity Talk non-completers

SUMMARY:
Dying patients and their families face many challenges near the end-of-life. Not only do patients often experience physical distress, but they also have feelings of loss of dignity, isolation, and uncertainty. Family members also face many challenges. They bear witness to the suffering of loved ones, and they face uncertainty, loss, and at times a mounting sense of helplessness.

The purpose of this study is to introduce and evaluate a new intervention called Dignity Talk, meant to enhance end-of-life experience for both patients and their families. Dignity Talk is based on a set of questions by which terminally ill patients and their family members can engage in meaningful conversations with each other. It is intended to lessen feelings of loss and helplessness and enhance feelings of connectedness by facilitating conversations that tap into a sense of meaning and purpose, sharing of memories, wishes, hopes, and giving guidance to those who will soon be left behind.

In Phase 1, 20 patients and family members will help finalize the method and Dignity Talk question framework (is it easy to understand, do the investigators have the right questions, and is the wording sensitive). In Phase 2 of the study the investigators will ask 100 patient-family pairs for feedback about Dignity Talk: what influence it had on their palliative care experience, whether it works well, and whether this intervention should become a regular part of palliative care. The investigators will also ask for feedback from health-care providers in both phases. We are requesting approval for an amendment to the healthcare provider feedback focus group questions. Will add those documents when they are approved.

Four to six months after the death of their loved one, the investigators will contact the family member to ask their thoughts about Dignity Talk, how it shaped their experience of their grief and bereavement.

The investigators expect that the study will show that Dignity Talk can be an effective, highly accessible palliative care intervention, which will enhance the end-of-life experience for palliative patients and the families who support them.

DETAILED DESCRIPTION:
See above summary

ELIGIBILITY:
Inclusion Criteria:

For Patient:

Patients being cared for:

* in a palliative care unit or whose care is focused on palliation as determined by clinical staff
* or patients who have have a confirmed diagnosis of amyotropic lateral sclerosis, and have symptoms in a domain that interferes with their social or occupation functioning: a) mobility, b) dysphasia, c) dyspnea, or d) speech or patients who have are have been on dialysis > 3 months and are > 60 years of age - or residents of Personal Care Home all of whom are:
* 18 years of age or older
* able to provide informed oral and written consent
* cognitive capacity (based on clinical consensus)

For Family Member or Close Friend:

* Family member or close friend who the patient identifies they would be comfortable talking with using the Dignity Talk question framework
* Family member who is 18 years of age or older
* Family member who is able to provide oral and written consent
* Family member who has cognitive capacity to participate in meaningful conversation (based on research staff decision)

For Healthcare Provider:

* Employed one of the participating sites
* in a discipline directly involved in clinical care (physician, nursing, social work, spiritual care, allied healthcare, etc.)

Exclusion Criteria:

* not meeting the above inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Family communication connectedness Index | 31 months

SECONDARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 31 months

CONTACTS AND LOCATIONS:
Locations (13):
- Canada (13):
  - Victoria Hospice, Victoria, British Columbia
  - St. Boniface Hospital, Winnipeg, Manitoba
  - Riverview Health Centre, Winnipeg, Manitoba
  - Concordia Hospital, Winnipeg, Manitoba
  - Deer Lodge Centre, Winnipeg, Manitoba
  - Grace Hospital, Winnipeg, Manitoba
  - Health Sciences Centre, Winnipeg, Manitoba
  - Manitoba Renal Program, Winnipeg, Manitoba
  - Seven Oaks Hospital, Winnipeg, Manitoba
  - Victoria Hospital, Winnipeg, Manitoba
  - Winnipeg Regional Health Authority, Winnipeg, Manitoba
  - WRHA Personal Care Homes, Winnipeg, Manitoba
  - Dr. Bob Kemp Hospice, Hamilton, Ontario

REFERENCES:
- [Derived] Guo Q, Chochinov HM, McClement S, Thompson G, Hack T. Development and evaluation of the Dignity Talk question framework for palliative patients and their families: A mixed-methods study. Palliat Med. 2018 Jan;32(1):195-205. doi: 10.1177/0269216317734696. Epub 2017 Nov 13. PMID 29130367